CLINICAL TRIAL: NCT02767011
Title: Tele-Health Electronic Monitoring to Reduce Post Discharge Complications and Surgical Site Infections Following Arterial Revascularization With Groin Incision
Brief Title: Tele-Health Electronic Monitoring to Reduce Post Discharge Complications and Surgical Site Infections
Acronym: THEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CAMC Health System (Other)
Collaborators: WVCTSI (Unknown)
Responsible Party: Principal Investigator, Albeir Mousa, Albeir Mousa MD, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-169
Record Dates: First submitted 2016-05-05; First posted 2016-05-10 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Peripheral Vascular Disease
Keywords: surgical site infection
MeSH Terms: conditions — Peripheral Vascular Diseases; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- THEM (Experimental): Patients receive telehealth electronic health care monitoring.
  Interventions: Other: Tele-Health Electronic Monitoring (THEM)
- Standard of Care (SOC) (No Intervention): Patients receive normal standard of follow-up care

INTERVENTIONS:
Other: Tele-Health Electronic Monitoring (THEM) — Patients in the intervention group (THEM) will receive a tablet computer and home monitoring medical devices with sensors to transmit the information to a central website that will be monitored by care managers. Medical devices will include weight scales, blood pressure cuffs and blood glucometers. Clinical care mangers will remotely monitor the patients and all electronic readings. Clinical care managers will call or send text messages to the patients based on alerts generated by the tele-health monitoring system.
  Arms: THEM

SUMMARY:
Abstract:

It is intuitive that post discharge surgical complications are associated with increased patient dissatisfaction, and directly associated with an increase in medical expenditures. It is also easy to make the connection that many post hospital discharge surgical complications including surgical site infections could be influenced or exacerbated by patient co-morbidities. The authors of a recent study reported that female gender, obesity, diabetes, smoking, hypertension, coronary artery disease, critical limb ischemia, chronic obstructive pulmonary disease, dyspnea, and neurologic disease were all of among significant predictors of surgical site infections after vascular reconstruction was performed. The main concern for optimal patient care especially in geographically isolated areas of West Virginia is to have early, expeditious, and prompt diagnosis of early surgical site infection with subsequent indicated interventions. This theme will lead to patient satisfaction, minimizing third party interventions and decrease the total cost associated with these complications. Nevertheless, it seems reasonable to believe that monitoring using telehealth technology and managing the general health care patients receive after a hospital vascular intervention will improve overall health and reduce post-operative complications.

Aims/Objectives:

1. The primary objective of the current project is to compare early and late outcomes for patients who receive post discharge health care monitoring (which includes using Telehealth electronic monitoring; THEM) to patients who receive standard of care (SOC) and routine discharge instructions and no monitoring.

Methods:

1. Randomize patients who are scheduled to have revascularization interventions with groin incisions to receive either telehealth electronic health care monitoring or normal standard of follow-up care.
2. Follow patients for 4 weeks, record any 30-day hospital readmissions or complications. In addition, have participants complete the follow-up survey questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with any planned vascular procedures with cut-down access to the groin and treated by one of the Charleston Area Medical Center -Vascular Surgeons in the Vascular Center (VCOE) will be consented and enrolled.

Exclusion Criteria:

1. do not plan to do follow-up visit at the VCOE;
2. history of dementia;
3. do not have home internet service with WIFI or live outside of the provided cell coverage area (cell coverage will be provided for patients without internet WIFI).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mousa AY, Broce M, Davis E, McKee B, Yacoub M. Telehealth electronic monitoring to reduce postdischarge complications and surgical site infections after arterial revascularization with groin incision. J Vasc Surg. 2017 Dec;66(6):1902-1908. doi: 10.1016/j.jvs.2017.07.063. PMID 29169546

RESULTS

PARTICIPANT FLOW:
Groups:
- THEM: Intervention Group. Received Tele-health monitoring
- Control: Control Group (received standard of care)
Period: Overall Study
Arm/Group | THEM | Control
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | THEM | Control | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (7.2) | 65.7 (7.3) | 64.0 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 10 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 16 | 13 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (4.3) | 29.1 (7.1) | 28.3 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: 30-Day Readmission (Any)
Description: Yes/No was patient readmitted? Patients were monitored for 30 days to see if they were re-admitted to the hospital for any reason. Percentage of patients with 30-day readmission.
Time Frame: 30-day
Measure: Count of Participants; unit: Participants
Arm/Group | THEM | Control
Number analyzed (Participants) | 16 | 14
Participants | 4 | 2

2. Primary Outcome: 30-day Wound Readmission
Description: Yes/No was patient readmitted for wound infection? Patients were monitored for 30 days to see if they were re-admitted to the hospital for wound infection. Percentage of patients with 30-day readmission for wound infection.
Time Frame: 30-day
Measure: Count of Participants; unit: Participants
Arm/Group | THEM | Control
Number analyzed (Participants) | 16 | 14
Participants | 1 | 1

3. Primary Outcome: Access Site/Wound Infections.
Description: Yes/No did patient any access site or would infections? Access site wounds for the patients were monitored for 30 days for any wound infections.
Time Frame: 30-day
Population: Percentage of patients with access site infections.
Measure: Count of Participants; unit: Participants
Arm/Group | THEM | Control
Number analyzed (Participants) | 16 | 14
Participants | 5 | 1

4. Secondary Outcome: The Difference Between Baseline and 30-day Quality of Life (Short-Form 8) Physical Summary Score
Description: The Difference between baseline and 30-day quality of life (Short-Form 8) Physical summary T-scores. The short-form (SF-8) Health Survey is an 8-item survey designed to measure quality of life. The SF-8 has 8 questions that first measures eight ordinal items (i.e., 1-5 Likert scale): general health, physical health functioning, role physical, bodily pain, vitality, social functioning, mental health and emotional roles. Summing the responses of the 8 items can be used to report an overall measure of physical and mental functioning. The raw Likert scale scores are converted to normalized standard T scores with a mean of 50 and standard deviation of 10. Measuring physical and mental health both before and after an intervention, as continuous summary scores can indicate better self-reported quality of life with higher scores. A difference score of 0 would indicate no change, while a larger positive difference score would indicate an increase in self-reported quality of life.
Time Frame: 30-day
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | THEM | Control
Number analyzed (Participants) | 16 | 14
T-scores
  Baseline Physical Summary Score | 27.76 (7.38) | 30.14 (11.28)
  30-day Physical Summary Score | 36.83 (8.58) | 34.61 (10.69)
  Difference (30-day - baseline) Summary Score | 9.07 (6.02) | 4.47 (7.63)

5. Secondary Outcome: Patient Satisfaction as Measured by the General Satisfaction Sub-scale of the Short-Form Patient Satisfaction Questionnaire (PSQ18)
Description: Patients' satisfaction was compared using the General Satisfaction sub-scale of the Short-Form Patient Satisfaction Questionnaire (PSQ18). The PSQ-18 contains 18 items (questions) that can measure seven dimensions of satisfaction: general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, and accessibility and convenience. Responses to the PSQ-18 require a selection on a Likert scale from 1 Strongly Agree to 5 Strongly Disagree with some of the questions worded in such a manner that agreement reflects greater satisfaction (1, 2, 3, 5, 6, 8, 11, 15 & 18). These responses were "re-coded" in order for a larger number to reflect greater satisfaction. Next, two individual items (3 and 17) are summed and averaged to produce the general satisfaction sub-scale. A larger number reflects greater satisfaction, with a range of 1 to 5.
Time Frame: 30-day
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | THEM | Control
Number analyzed (Participants) | 16 | 14
units on a scale | 4.0 [4.0 to 4.5] | 3.75 [2.87 to 4.5]

6. Secondary Outcome: Number of Participants With Home Nursing Visits
Description: Yes/No did the patient have (any) home nursing visits during the 30-day follow-up period.
Time Frame: 30-day
Measure: Count of Participants; unit: Participants
Arm/Group | THEM | Control
Number analyzed (Participants) | 16 | 14
Participants | 3 | 3

7. Secondary Outcome: Stroke
Description: Yes/No did patient have a stroke. Patients were monitored for 30 days for stroke.
Time Frame: 30-day
Measure: Count of Participants; unit: Participants
Arm/Group | THEM | Control
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

8. Secondary Outcome: Myocardial Infarction
Description: Yes/No did patient have myocardial infarction. Patients were monitored for 30 days for myocardial infarction.
Time Frame: 30-day
Measure: Count of Participants; unit: Participants
Arm/Group | THEM | Control
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

9. Secondary Outcome: Death
Description: Yes/No Did patient die? Patients for monitored for 30 days for death.
Time Frame: 30-day
Measure: Count of Participants; unit: Participants
Arm/Group | THEM | Control
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients were monitored for 30 days for any adverse events.
Arm/Group | THEM | Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT02767011/Prot_SAP_000.pdf